CLINICAL TRIAL: NCT03543215
Title: Can Staging Magnetic Resonance Imaging (MRI) Features Prognosticate Patients Presenting With Endometrial Cancer?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 16HH3687 Radiomics EC
Record Dates: First submitted 2017-06-30; First posted 2018-06-01 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Endometrial Cancer; Endometrial Neoplasms
Keywords: MRI; Radiomics; Texture features; Prognostication; Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Radiomics: Analysis of textural features of imaging (MRI and Ultrasound) — All patients with confirmed endometrial cancer will have received Ultrasound and MRI as part of routine standard of care. Textural features from this will be analysed to see if can predict prognosis.

SUMMARY:
Aim: Assess the value of MRI features in predicting prognosis in patients with endometrial cancer

This study will examine the MRI features of women with confirmed endometrial cancer to see if textural features can prognosticate patients.

DETAILED DESCRIPTION:
Aim: Assess the value of MRI features in predicting prognosis in patients with endometrial cancer

Background:

Endometrial cancer is the commonest gynaecological cancer in the United Kingdom. MR Imaging is used to provide pre-treatment local staging in Endometrial Cancer based on the FIGO staging system. This MRI stage is used by clinicians, in combination with pre-operative histology and clinical assessment of the patient, to counsel patients about their prognosis.

Currently the information obtained from the MRI study is largely anatomical and concerns the extent of local tumour spread at the time of diagnosis. Each stage under the FIGO system is associated with a prognosis based on data from the literature. Important prognostic indicators include the depth of tumour invasion in the uterine muscle (myometrium), invasion of the cervical stroma by tumour, spread to lymph node tissues and the histological sub-type of tumour present.

However, with ever improving MRI technology there are now newer sequences employed as part of the staging study which may potentially yield more information. In other cancer types, e.g. prostate, breast and liver, textural analysis of the tumour on pre-treatment imaging (CT/PET-CT/MRI) is being analysed to try and identify features which could be used as prognostic markers for patient outcome.

The Study:

All patients with confirmed cancer on histology will receive an Ultrasound and MRI as part of routine care. The MRI scan will include T1, T2, DWI and contrast enhanced sequences. Patients referred to Hammersmith Hospital from other trusts who are diagnosed with endometrial cancer will be approached for consent and enrolment into latter part of study. These patients will have had an MRI but may not have had all the sequences needed and may therefore require a further MRI scan with additional sequences. These images will be saved and analysed. Pathological findings (e.g. type and grade of cancer) will be correlated with the radiological results.

Definitive management of endometrial cancer includes a hysterectomy for most patients. Following surgery patients will continue with routine standard of care and follow up. Patients will be followed up for 5 years to provide 5 year survival data. Images from ultrasound and MRI pelvis will be analysed to see if they can predict the 5 year survival.

This prospective study will also be used to validate a retrospective model using MRI textural features in endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* All women presenting with a confirmed diagnosis of endometrial cancer
* Reviewed at the Specialist Gynaecology Oncology MDT
* Have MR Imaging and Hysterectomy specimens available for review.

Exclusion criteria:

* Anyone lacking capacity.
* <18years old.
* Pregnant.
* No MR Imaging available for review -- No pathology specimen available for review

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is on endometrial cancer
Study Population: All patients reviewed at the Specialist Gynaecology Oncology MDT at ICHNT with a diagnosis of endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
To assess the value of MRI features in predicting prognosis in patients with endometrial cancer using progression free survival (PFS) and overall survival (OS) as end points | 8 years (3 year data collection and 5 year follow up).
  Assess features of pelvic MRIs (including (i) tumour image intensity, (II) shape, (III) texture and (IV) multiscale wavelet) and create a mathematical algorithm to predict prognostic outcome (5 year survival).

SECONDARY OUTCOMES:
Assess the correlation between imaging features and histopathological features. | 3 years
  Assess textural features of pelvic MRI in conjunction with histopathology (type of tumour, grade LVSI, 'aggressiveness' of cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Charlotte and Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Marcus D, Russell J, Aboagye EO, Ellis LB, Sheeka A, Park WE, Bharwani N, Ghaem-Maghami S, Rockall AG. Weibull parametric model for survival analysis in women with endometrial cancer using clinical and T2-weighted MRI radiomic features. BMC Med Res Methodol. 2024 May 9;24(1):107. doi: 10.1186/s12874-024-02234-1. PMID 38724889